CLINICAL TRIAL: NCT06981429
Title: A Positive Food Parenting Intervention to Promote Healthy Growth in Children at Risk for Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katherine Balantekin, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00008522; R03DK138232 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Obesity; Nutrition Disorder
Keywords: children; parenting; parent feeding practices; food parenting; obesity risk; positive food parenting; autonomy promotion; structure - based food parenting
MeSH Terms: conditions — Pediatric Obesity; Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Participants will either be assigned to the control group or the experimental group. The control group will participate in a 10 - session 'promoting healthy development in middle childhood' program. The experimental group will be receiving the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Positive Food Parenting Intervention (Experimental): Participants randomly assigned to the experimental group.
  Interventions: Behavioral: Nourish to Flourish: The Power of Positive Food Parenting
- Control Group (No Intervention): Participants randomly assigned to the control group.

INTERVENTIONS:
Behavioral: Nourish to Flourish: The Power of Positive Food Parenting — This intervention focuses on increasing diet quality and parent use of positive food parenting practices with the goal of promoting healthy child growth). This will be a 12 - week, 12 session study. Sessions 1 and 12 will consist of collection baseline and post-intervention data. Sessions 2 - 11 will be a mix of online - group sessions and individual online or in - person sessions (based on participant preference). The group sessions are focused on principal investigator presentation of the intervention curriculum and group discussion. The individual sessions are focused on goal setting, coping planning, and working through individual situations with a trained coach.
  Arms: Experimental Group - Positive Food Parenting Intervention

SUMMARY:
This study is the pilot of a 12 - week positive food parenting intervention focused on structure-based and autonomy promoting practices. The intervention aims to give parents the tools to promote healthy child growth and improve diet quality. The investigators are piloting to assess feasibility and efficacy of the intervention through examining participant retention, impact on parent feeding practices, and impact on parent and child diet quality.

ELIGIBILITY:
PARENT CRITERIA:

Inclusion Criteria:

* Age > 18 years old.
* Have a child between the ages of 5 - 11 who is at risk for obesity (child BMI percentile > 85th) or parent it concerned about their child developing overweight or obesity
* Low use of positive food parenting (Defined as: low reports of individual nutrition education/ knowledge OR reports low levels of structure, involvement, or encouragement in their food parenting practices)
* Must be responsible for feeding their eligible child at least 50% of the time.
* Fluent in English.
* Have access to internet and a Zoom compatible device.

Exclusion Criteria:

* Age is < 18 years old. Their child is determined ineligible (based on BMI percentile and age).
* Does not report low use of positive food parenting (as defined above).
* Is responsible for feeding their eligible child < 50% of the time.
* Not fluent in English.
* Does not have access to internet and a Zoom compatible device.
* On medication that could influence their eating or feeding behaviors.

CHILD CRITERIA:

Inclusion Criteria:

* Their parent/ guardian is eligible and participating in the study.
* Ages 5 - 11
* Is not current diagnosed with a clinical eating disorder (ED).
* Is not on any medications, or have any conditions, that could influence the child's taste, appetite, or olfactory sensory responsiveness.

Exclusion Criteria:

* Their parent/ guardian is not eligible nor participating in the study.
* Below the age of 5 and above the age of 11.
* BMI percentile < 85th and/or > 97th.
* Current diagnosis of a clinical eating disorder (ED)
* Medications or conditions that could influence the child's taste, appetite, or olfactory sensory responsiveness.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Parent use of structure - based and autonomy - promoting parent feeding practices. | Session 1 (week 1) to Session 12 (week 12)
  Compare responses to validated questionnaires measuring food parenting practices from session 1 to session 12.
Parent and Child Diet Quality | Session 1 (week 1) and Session 12 (week 12)
  Compare change in parent and child healthy eating index (HEI) from session 1 to session 12. The healthy eating index (HEI) is a measure of how a participants diet aligns with the recommendations by the Dietary Guidelines for Americans (Dietary Guidelines). Possible scores range from 0 (does not align at all with recommendations by the Dietary Guidelines for Americans) to 100 (perfectly aligns with recommendations by the Dietary Guidelines for Americans). Higher scores mean a better outcome.
Parent BMI and Child zBMI | Session 1 (week 1) and Session 12 (week 12)
  Change in parent BMI and child zBMI from session 1 to session 12.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine N Balantekin, PhD, RD, Principal Investigator — Assistant Professor, University at Buffalo
Locations (1):
- State University of New York at Buffalo, South Campus, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided